CLINICAL TRIAL: NCT00226057
Title: Efalizumab for Moderate to Severe Atopic Dermatitis - A Phase I Pilot Study in Adults
Brief Title: Efalizumab for Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Eric Simpson, M.D., M.C.R., Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 578
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic dermatitis; Raptiva
MeSH Terms: conditions — Dermatitis, Atopic | interventions — efalizumab

ARMS (1):
- Raptiva Open Label (Experimental): Raptiva administered by weekly subcutaneous injections. First dose of 0.7mg/kg. Subsequent doses will be of 1mg/kg SQ weekly.
  Interventions: Drug: Raptiva

INTERVENTIONS:
Drug: Raptiva — Open Label
  Other Names: Efalizumab

SUMMARY:
The purpose of this study is to determine if Raptiva will have beneficial effects in the treatment of patients with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis is a common, highly pruritic, inflammatory skin disease that affects up to 17% of school-aged children. Most cases of childhood atopic dermatitis improve or resolve by adulthood. However, the majority of patients retain some features of atopic dermatitis and some continue to have severe disease that continues to adulthood. Moderate to severe atopic dermatitis cannot be adeuately controlled with topical agents. Consequently many patients are treated with systemic corticosteroids, cyclosporine, azathioprine, methotrexate, and other immunosuppressants that carry the risk of severe atopic dermatitis is greatly needed. The chronic use of current immunosuppressive agents is limited by cumulative end-organ toxicities. We propose inhibition of T cell trafficking to the skin with Raptiva will have beneficial effects in the treatment of patients with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age >= 18 years
* If a female of child bearing potential, a negative pregnancy test and commitment to birth control for the duration of the study are necessary.
* Diagnosis of atopic dermatitis using the Hanifin-Rajka criteria
* Disease severity of Moderate or Severe on the Rajka-Langeland Severity Score
* Candidate for, or previously on systemic therapy, including cyclosporine, methotrexate, ultraviolet light or other immunosuppressant. Specifically, patients are considered candidates for systemic therapy when their disease is not adequately controlled using topical therapies or side-effects prevent the further safe use of topical therapies.
* Patients must meet the following washout requirements:

Pre-Study and Concomitant Washout Period Restriction (Baseline Therapy Restrictions Prior to Study Thru End of Study)

Investigational Drugs 4 Weeks Disallowed Light Treatments 4 Weeks Disallowed Systemic corticosteroid used 4 Weeks Disallowed for atopic dermatitis flare Topical tacrolimus or 2 Weeks Disallowed pimecrolimus Topical corticosteroids Must be on stable Allowed at stable doses dose for 2 weeks (Triamcinolone ointment 0.1% only) Any systemic 4 Weeks Disallowed immunosuppressive medication Topical and systemic antibiotics Cannot be on Allowed if infection antibiotics at the develops start of study

Exclusion Criteria:

* Patient's with known hypersensitivity to Raptiva (efalizumab) or any of its components
* Pregnant or lactating women
* Patients receiving immunosuppressive agents
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Participation in another simultaneous medical investigation or trial
* Subjects known to be immunocompromised(lymphoma, HIV+, Wiskott-Aldrich syndrome)
* Systemic corticosteroid-dependent asthma
* Active infection of any type at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2005-11 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and effectiveness of Raptiva in patients with moderate to severe atopic dermatitis | EASI Score collected at 12 weeks following baseline
  The primary efficacy outcome measure will be the change in mean Eczema Area and Severity Index (EASI) score from baseline

SECONDARY OUTCOMES:
Improvement in EASI score | Assessed 12 weeks after baseline
  Total percent of patients reaching 50% improvement in EASI score
Improvement in IGA score | Assessed 12 weeks after baseline
  Numbers of patient reaching clear, almost clear or mild disease on the Investigator Global Assessment (IGA) Score
Subject's assessment of overall response | End of study
  Subject's assessment of overall response
Change in serum IgE level | Serum IgE collected at 12 weeks following baseline
  Change in serum IgE Level
Pruritis (0-10 VAS Scale) change | VAS scale collected at 12 weeks following baseline
  Pruritis (0-10 VAS Scale) change
Time to first response | Assessed on Days 28,56, and 84
  Time to first response as defined by a decrease of 25% in EASI score

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Simpson, MD, Principal Investigator — Oregon Health and Science University

REFERENCES:
- [Background] Laughter D, Istvan JA, Tofte SJ, Hanifin JM. The prevalence of atopic dermatitis in Oregon schoolchildren. J Am Acad Dermatol. 2000 Oct;43(4):649-55. doi: 10.1067/mjd.2000.107773. PMID 11004621
- [Background] Williams HC, Strachan DP. The natural history of childhood eczema: observations from the British 1958 birth cohort study. Br J Dermatol. 1998 Nov;139(5):834-9. doi: 10.1046/j.1365-2133.1998.02509.x. PMID 9892950
- [Background] Werther WA, Gonzalez TN, O'Connor SJ, McCabe S, Chan B, Hotaling T, Champe M, Fox JA, Jardieu PM, Berman PW, Presta LG. Humanization of an anti-lymphocyte function-associated antigen (LFA)-1 monoclonal antibody and reengineering of the humanized antibody for binding to rhesus LFA-1. J Immunol. 1996 Dec 1;157(11):4986-95. PMID 8943405
- [Background] Leung DY, Bhan AK, Schneeberger EE, Geha RS. Characterization of the mononuclear cell infiltrate in atopic dermatitis using monoclonal antibodies. J Allergy Clin Immunol. 1983 Jan;71(1 Pt 1):47-56. doi: 10.1016/0091-6749(83)90546-8. PMID 6337197
- [Background] Reitamo S, Wollenberg A, Schopf E, Perrot JL, Marks R, Ruzicka T, Christophers E, Kapp A, Lahfa M, Rubins A, Jablonska S, Rustin M. Safety and efficacy of 1 year of tacrolimus ointment monotherapy in adults with atopic dermatitis. The European Tacrolimus Ointment Study Group. Arch Dermatol. 2000 Aug;136(8):999-1006. doi: 10.1001/archderm.136.8.999. PMID 10926735
- [Background] Hanifin JM, Schneider LC, Leung DY, Ellis CN, Jaffe HS, Izu AE, Bucalo LR, Hirabayashi SE, Tofte SJ, Cantu-Gonzales G, et al. Recombinant interferon gamma therapy for atopic dermatitis. J Am Acad Dermatol. 1993 Feb;28(2 Pt 1):189-97. doi: 10.1016/0190-9622(93)70026-p. PMID 8432915